CLINICAL TRIAL: NCT01031576
Title: Postural Analysis and Eletromiographic Activity in Patients With Knee Osteoarthritis
Brief Title: Postural Analysis in Patients With Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: POSTURAL ANALYSIS AND ELETROMIOGRAPHIC ACTIVITY IN PATIENTS WITH KNEE OSTEOARTHRITIS, University of Sao Paulo
Other Study IDs: 12345
Record Dates: First submitted 2008-04-02; First posted 2009-12-14 (Estimated); Last update posted 2009-12-14 (Estimated); Status verified 2008-04

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis, posture, knee
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Osteoarthritis is the result of the degeneration of the cartilage to articulate, being currently considered as having an multifactorial cause.The knees are one of the affected joints more due to overload that constitutes the main activator or determinative mechanism for the development of the illness. Beyond pain it has important reduction of the amplitude of movement and the muscular force that causes functional limitation and posture's alterations intervening with the activities of daily life. Therefore, the main objective of this study will be to characterize the posture's alterations and the electromiographic activity in patients with osteoarthritis of knees. For this study 30 citizens will be evaluated, 15 with diagnosis of OA of knees unilaterally and 15 healthful citizens, both the groups will be of the feminine sex with age between 60 to 80 years. The selected patients will answer a questionnaire of personal dates and will have an evaluation fiche, in which will be written down: age, index of corporal mass (IMC), index of Lesquene, index WOMAC (Western Ontario and Mac Master), personal and familiar date of the diagnosis, antecedents, instituted treatments, date of the last x-ray, radiological classification of the osteoarthritis according to Scale of Kellgren, electromiographics date and seeming of the postural evaluation. For the electromiographic evaluation the activity of the muscles vastus lateralis and medial oblique in the isometric contraction maximum volunteer (ICMV) and in the march will be analyzed. And for the postural evaluation will be made three photographs in the sights previous frontal and sagittal right and left, being that, for the analysis of the posturais alterations the program will be used SAPO.

DETAILED DESCRIPTION:
Osteoarthritis is the result of the degeneration of the cartilage to articulate, being currently considered as having an multifactorial cause. Of the histological point of view it is characterized for alterations of the loss of the natural viscoelasticity, giving to origin the foci of "softening" in the cartilaginous surface that if gets depressed becoming discontinues for the appearance of "fibrillation zones" provoking reaction of the subcondral bone that if condemns in the pressure areas (sclerosis) and proliferates together to the edges of the joint (osteophytic). It is that affect millions of people annually and one of the main and a common condition causes pain functional incapacity generating enormous economic load for the community. The knees are one of the affected joints more due to overload that constitutes the main activator or determinative mechanism for the development of the illness. Beyond pain it has important reduction of the amplitude of movement and the muscular force that causes functional limitation and posture's alterations intervening with the activities of daily life. Therefore, the main objective of this study will be to characterize the posture's alterations and the electromiographic activity in patients with osteoarthritis of knees. For this study 60 citizens will be evaluated, 30 with diagnosis of OA of knees unilaterally and 30 healthful citizens, both the groups will be of the feminine sex with age between 65 to 75 years. The selected patients will answer a questionnaire of personal dates and will have an evaluation fiche, in which will be written down: age, index of corporal mass (IMC), index of Lesquene, index WOMAC (Western Ontario and Mac Master), personal and familiar date of the diagnosis, antecedents, instituted treatments, date of the last x-ray, radiological classification of the osteoarthritis according to Scale of Kellgren, electromiographics date and seeming of the postural evaluation. For the electromiographic evaluation the activity of the muscles vastus lateralis and medial oblique in the isometric contraction maximum volunteer (ICMV) and in the march will be analyzed. And for the postural evaluation will be made three photographs in the sights previous frontal and sagittal right and left, being that, for the analysis of the posturais alterations the program will be used SAPO (software for postural evaluation - version 0.63).

In the analysis descriptive statistics the average, medium and shunting line will be used standard. The level of significance will be established in α < 0,05.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Osteoarthritis Disease

Exclusion Criteria:

* Others Disease orthopedics

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 15 with diagnosis of OA of knees unilaterally and 15 healthful citizens, both the groups will be of the feminine sex with age between 65 to 75 years
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2006-02; Primary Completion 2008-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luciano Sencovici, Principal Investigator — USP
Locations (1):
- Luciano Sencovici, São Paulo, São Paulo, Brazil